CLINICAL TRIAL: NCT01678612
Title: Efficacy of Copper in Reducing Health-Acquired Infections and Microbial Burden as Measured on High Touch Surfaces in a Pediatric Intensive Care Unit. A Controlled Clinical Trial.
Brief Title: Efficacy of Copper in Reducing Health-Acquired Infections in a Pediatric Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Codelco (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CODEHRdR
Record Dates: First submitted 2012-08-25; First posted 2012-09-05 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Nosocomial Infections
Keywords: Copper; Health-Acquired Infections; Bacterial Load; Intensive Care Units, Pediatric
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non copper standard surfaced objects (No Intervention): Rooms assigned to standard surfaced objects
- Copper-alloy surfaced objects (Experimental): Rooms furnished with copper surfaced objects, i.e. bed rails, bed rail levers, IV poles, nurse workstation, clipboards, sink handles.
  Interventions: Other: Copper-alloy surfaced objects

INTERVENTIONS:
Other: Copper-alloy surfaced objects — Room assigned to the Experimental arm will be furnished with copper-alloy surfaced objects,i.e. bed-rails, bed-rail levers, IV poles, nurse workstation, HCW clipboards, sink handles.
  Arms: Copper-alloy surfaced objects

SUMMARY:
Healthcare-acquired infections (HAI) cause substantial patient morbidity and mortality. Commonly touched items in the patient care environment harbor microorganisms that may contribute to HAI risk. The purpose of this study is to assess whether placement of copper-alloy surfaced objects in a pediatric intensive care unit (PICU) reduce risk of HAI in comparison with non-copper surfaced objects.

ELIGIBILITY:
Inclusion Criteria:

* patient admitted to PICU
* stay at PICU > 24 hours
* informed consent by parent/legal representative

Exclusion criteria: none

Ages: 7 Days to 180 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1012 (Actual)
Dates: Start 2012-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Hospital-Acquired Infections (HAI) incidence density / 1,000 patient-days | Participants will be followed for the duration of hospital stay, an expected average of 6 days

SECONDARY OUTCOMES:
Microbial Burden measured on high-touch copper and non-copper surfaced objects | 1 year study duration
  Total microbial burden and selected bacteria (MRSA,VRE) will be measured twice a month in all bedrails and sink handles of the PICU study site.

OTHER OUTCOMES:
Incidence of new events of colonization with selected pathogens per 1000 patient-days at risk | participants will be followed for the duration of hospital stay, an expected average of 6 days
  Patients with negative culture (from skin and mucosa samples) will be sampled at Day 3, Day 6 and discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Bettina von Dessauer, MD, Principal Investigator — Hospital Roberto del Rio
Locations (1):
- Hospital Roberto del Rio, Santiago, Chile